CLINICAL TRIAL: NCT07221981
Title: Clinical and dEmographic chaRacteristics of Patients With Frequent COPD Exacerbations and Evaluation of Therapeutic Approaches in Treatment in RussiA
Brief Title: Study of Patient With Frequent COPD Exacerbations
Acronym: CERERA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00123
Record Dates: First submitted 2025-05-13; First posted 2025-10-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Study is a multicenter, non-interventional, observational, ambispective (retrospective-prospective) study to evaluate clinical and demographic characteristics, approaches to therapy in outpatients with COPD and frequent exacerbations in the Russian Federation. Planned number of Study site is 35 outpatient centers with experience of treatment of COPD with frequency exacerbations in about 30 regions in Russia.

DETAILED DESCRIPTION:
The study consists of a retrospective phase covering 52 weeks and a prospective phase of 24 weeks, involving 2000 patients across approximately 35 cites. Therefore, the aim of the study is to evaluate the clinical and demographic patients' characteristics based on retrospective part and COPD treatment patterns based on prospective part of patients with frequent exacerbations of COPD on dual therapy in the Russian Federation. The study results will be interpreted in the context of an open label, single arm study design. Due to the limited data available on the COPD population in Russia, the characterization of clinical and demographic characteristic of patients based on the retrospective component of the study will enhance the understanding of this patient group and the prospective aspect, which analyses therapeutic approaches, will help to assess physicians' adherence to current recommendations regarding therapy selection for COPD patients on dual therapy with frequent exacerbations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of inclusion;
2. Signed and dated written informed consent in accordance with ICH-GCP and local law prior to inclusion in the study;
3. Patients with diagnosed moderate-to-severe COPD (see comments below);
4. ≥2 moderate or ≥1 severe COPD exacerbations in previous 52 weeks (see comments below);
5. Patients have been receiving two inhaled maintenance therapies (LABA/LAMA, ICS/LABA, ICS/LAMA) for at least 6 weeks prior to inclusion.

Exclusion Criteria:

1. Current or previous treatment with triple combination (ICS/LABA/LAMA) within 52 weeks prior to inclusion;
2. COPD due to documented α-1 antitrypsin deficiency;
3. A diagnosis of bronchiectasis, sarcoidosis, interstitial lung diseases, or idiopathic pulmonary fibrosis, exacerbation of bronchial asthma or any acute or chronic disease that, as deemed by Investigator, limits the ability of patients to participate in this study or could influence the interpretation of the results;
4. The participation in any clinical study currently or within 52 weeks prior to inclusion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2000 adult patients with diagnosed moderate-to-severe COPD and ≥2 moderate or ≥1 severe exacerbations in previous 52 weeks despite two inhaled maintenance therapies (LABA/LAMA, ICS/LABA, ICS/LAMA) for at least 6 weeks prior to inclusion and are monitored and treated by pulmonologists or general practitioners
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To describe the baseline Demographic data characterisics of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Demographic data
  1. Mean age at the inclusion into the study, and age groups (<50; 50-65, >65 years);
  2. Mean age at the primary COPD diagnosis;
  3. Proportion of men and women;
  4. Proportion of patients with each educational status (higher, secondary special, secondary general) at inclusion;
  5. Proportion of patients from each residential region of Russia;
To describe the baseline Negative lifestyle factors characterisics of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Negative lifestyle factors 6. Proportion of patients with negative lifestyle factors at inclusion (evaluated on Visit 1 based on patient's interview):
  a. Proportion of patients with history of smoking (former smoker)/current smokers - applicable for tobacco and e-cigarettes (vapes) smoking; d. Proportion of patients with overeating; e. Proportion of patient with physical inactivity.
To describe the baseline Anthropometry data characterisics of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Anthropometry data 7. Mean body mass index (BMI) at inclusion (in previous 52 weeks (the most recent available value) or evaluated on Visit 1);
To describe the baseline COPD drug treatment duration in previous 52 weeks of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  9. Proportion of patients receiving different classes of drugs for treatment of COPD during prior 52 weeks before inclusion. The following classes of drug or their combinations will be collected. The combinations may be prescribed as separate drugs or fixed combination (of ≥1 drug class in one medication):
  1. SABA alone;
  2. ICS alone
  3. LABA alone
  4. LAMA alone
  5. LABA and LAMA
  6. ICS and LABA
  7. ICS and LAMA
  8. LABA and LAMA plus:
  a) Macrolide antibiotics b) CS
To describe the baseline Cardiovascular diseases of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Cardiovascular diseases 10. Proportion of patients with cardiovascular diseases (cardiac failure, ischaemic heart disease, myocardial infarction, arrhythmia, stroke) at inclusion (diagnosed in medical documentation ever or identified on the Visit 1 via a patient interview);
To describe the baseline other comorbidities of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Other comorbidities 11. Proportion of patients with different other comorbidities at inclusion (diagnosed in previous 52 weeks or on Visit 1);
To describe the baseline Blood eosinophils count of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Blood eosinophils count 12. Mean blood eosinophils count (cells/μl) at inclusion (in previous 52 weeks (the most recent available value) or evaluated on Visit 1); 13. Proportion of patients with different levels of blood eosinophils count at inclusion (in previous 52 weeks (the most recent available value) or evaluated on Visit 1):
  1. <150 cells/μl;
  2. ≥150 cells/μl;
  3. ≥300 cells/μl.
To describe the baseline mean smoking index . | 52 weeks of retrospective data before visit 1
  applicable for current/former tobacco smokers (pack-years)
To describe the baseline mean duration of smoking | 52 weeks of retrospective data before visit 1
  applicable for current/former e-cigarettes (vapes) smokers (years);
To describe the Proportion of patients with overweight | 52 weeks of retrospective data before visit 1
  determined as BMI ≥25 kg/m2 at inclusion (in previous 52 weeks (the most recent available value) or evaluated on Visit 1
To describe the baseline dosages of COPD drug treatment in previous 52 weeks of outpatients with moderate and severe COPD. | 52 weeks of retrospective data before visit 1
  Proportion of patients receiving different classes of drugs for treatment of COPD. The following classes of drug or their combinations will be collected. The combinations may be prescribed as separate drugs or fixed combination (of ≥1 drug class in one medication):
  1. dosage SABA alone ;
  2. dosage ICS alone
  3. dosage LABA alone
  4. dosage LAMA alone
  5. dosage LABA and LAMA
  6. dosage ICS and LABA
  7. dosage ICS and LAMA
  8. LABA and LAMA plus:
  a) dosage Macrolide antibiotics b) dosage CS

SECONDARY OUTCOMES:
To describe the proportion of patients receiving different classes of drugs for treatment of COPD between V1 and V2 | 24 weeks after visit 1
  the proportion of patients with prescribed of the following classes of drug or their combinations. The combinations may be prescribed as separate drugs or fixed combination (of ≥1 drug class in one medication):
  1. SABA alone
  2. LABA alone
  3. LAMA alone
  4. ICS alone
  5. ICS and LABA
  6. ICS and LAMA
  7. LABA and LAMA
  8. ICS and LABA and LAMA (triple therapy)
To describe Healthcare resource utilization during 24-week prospective study follow-up compared to baseline period | 24 weeks after visit 1
  7. Proportion of patients with healthcare resource utilization events due to COPD during 52 weeks prior to inclusion (Visit 1):
  * Unscheduled outpatient visits;
  * Emergency department visits/emergency calls;
  * Hospitalizations. 8. Proportion of patients with healthcare resource utilization events due to COPD occurred from inclusion (Visit 1) to Visit 2:
  * Unscheduled outpatient visits;
  * Emergency department visits/emergency calls;
  * Hospitalizations.
To describe changes of Mean forced expiratory volume during 24-week prospective study follow-up compared to baseline | 24 weeks after visit 1
  11. Mean parameters of lung function at inclusion (Visit 1) and Visit 2:
  a. Mean forced expiratory volume in 1 second (pre- and post-FEV1); 12. change from baseline (Visit 1) to Visit 2:
  a. Pre- and post-bronchodilator FEV1;
To describe Change in CAT score during 24-week prospective study follow-up compared to baseline | 24 weeks after visit 1
  13. Mean baseline in the COPD Assessment Test (CAT) score at inclusion; 14. Mean change from baseline (at inclusion) to 24 weeks (Visit 2) in the CAT score;
To describe Newly occurred cardiovascular diseases and other comorbidities during 24-week prospective study follow-up | 24 weeks after visit 1
  16. The proportion of patients with newly occurred cardiovascular diseases (cardiac failure, ischemic heart disease, myocardial infarction, arrhythmia, stroke) during study follow-up, the analysis includes withdrawn patients; 17. The proportion of patients with newly occurred other (non-cardiovascular) comorbidities during study follow-up, the analysis includes withdrawn patients.
To describe Blood eosinophils count during 24-week prospective study follow-up compared to baseline | 24 weeks after visit 1
  18. Mean blood eosinophils count (cells/μl) on Visit 2; 19. Proportion of patients with different levels of blood eosinophils count on Visit 2:
  1. <150 cells/μl;
  2. ≥150 cells/μl;
  3. ≥300 cells/μl. 20. Mean change in blood eosinophils count (cells/μl) from baseline (Visit 1) to Visit 2.
To describe COPD corticosteroid treatment during 24-week prospective study follow-up and change in therapy compared to baseline period | 24 weeks after visit 1
  3.Proportion of patients with CS prescribed during the study between Visit 1 and Visit 2 - overall and by type (CS intermittent; CS regularly);
To describe Proportion of patients with macrolide antibiotics during 24-week prospective study follow-up and change in therapy compared to baseline period | 24 weeks after visit 1
  prescribed during the study between Visit 1 and Visit 2.
To describe Proportion of patients with change of inhaled COPD therapy during the study during 24-week prospective study follow-up and change in therapy compared to baseline period | 24 weeks after visit 1
  between V1 and V2 compared to the baseline period (change in drug class: SABA alone, LABA alone, LAMA alone, ICS alone, open and fixed combination of ICS, LABA or LAMA, macrolide antibiotics; CS: intermittent or regularly; or starting of triple therapy with ICS/LABA/LAMA);
To describe Mean duration of COPD-related hospitalizations during 52 weeks prior to inclusion | 52 weeks of retrospective data before visit 1
  will be described at Visit 1
To describe Mean duration of COPD-related hospitalizations during 24-week prospective study follow-up compared to baseline period | 24 weeks after visit 1
  occurred from inclusion (Visit 1) to Visit 2.
To describe changes of Mean forced vital capacity during 24-week prospective study follow-up compared to baseline | 24 weeks after visit 1
  * Mean forced vital capacity (FVC) at Visit 1
  * Mean FVC change from baseline (Visit 1) to Visit 2
To describe changes of Mean post-bronchodilator FEV1/FVC ratio during 24-week prospective study follow-up compared to baseline | 24 weeks after visit 1
  * at Visit 1
  * change from baseline (Visit 1) to Visit 2
To describe Percent of responders using the CAT who achieved MCID (minimal clinically important difference) during 24-week prospective study follow-up compared to baseline | 24 weeks after visit 1
  Determined as 2 or more points after 24 weeks from baseline;
To describe Mean CS daily dose (mg/day in prednisolone equivalent) during the study between Visit 1 and Visit 2 during 24-week prospective study follow-up and change in therapy compared to baseline period | 24 weeks after visit 1
  evaluated in patients with CS prescribed during the study
To describe Proportion of patients with CS using for COPD exacerbations treatment during the study | 24 weeks after visit 1
  between Visit 1 and Visit 2 during 24-week prospective study follow-up and change in therapy dose compared to baseline period

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Research site, Ivanovo
  - Research site, Moscow
  - Research site "OOO Energy of health", Saint Petersburg
  - Research site, Saint Petersburg
  - Research site, Voronezh
  - Research site, Yekaterinburg